CLINICAL TRIAL: NCT00129740
Title: Therapy of Early Chronic Phase Chronic Myelogenous Leukemia (CML) With Oral Nilotinib
Brief Title: Phase II Nilotinib With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia (CML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0048; NCI-2012-01313 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Leukemia, Myelogenous, Chronic
Keywords: Chronic phase CML; Newly diagnosed chronic phase CML; AMN107
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental): 400 mg orally twice daily
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 400 mg orally twice daily
  Other Names: Tasigna®; AMN107

SUMMARY:
The goal of this clinical research study is to learn if an experimental agent, AMN107 (nilotinib), can help to control CML in chronic phase. The safety of this experimental agent will also be studied.

DETAILED DESCRIPTION:
Nilotinib is a drug that is designed to block a protein that is responsible for the development of CML.

If you are found to be eligible to take part in this study, you will take 2-4 nilotinib capsules or tablets by mouth 2 times a day (4-8 capsules or tablets a day total) every day, at least 8 hours apart. Nilotinib should be taken each morning and evening with a large glass of water. The study medication will be given to you every 3 - 12 months. You will also be given a "pill diary" to write down when (day and time) you take the drug. You will also write in the diary any side effects you may experience. You should bring the diary, any unused capsules or tablets, and empty containers of nilotinib with you to every visit to the study doctor. Any unused supplies must be returned at the end of the study.

Every 1-4 weeks during the first 4 weeks of the study, you will have around 2 teaspoons of blood drawn for routine blood tests. The blood tests will then be repeated every 4-8 weeks (or more often if your doctor feels it is necessary) until you have been on study for 6 months, then every 3 to 6 months for another 18 months. After that, you may have the blood tests repeated as often as the doctor thinks it is needed. A bone marrow sample will also be taken every 3-4 months for the first year and then every 6-12 months in the 2nd year, then every 2-3 years for as long as you are on the study to check on the status of the disease. Additionally, blood (about ½ tablespoon) will be drawn or a bone marrow sample will be collected every 3-4 months for the first year and then every 6-12 months until 2 years, and then about one time a year for as long as you are on the study to check on the status of the disease. However, if you are in complete remission after Year 2, your doctor will decide when you will have a bone marrow aspiration. But you will still have blood drawn (about ½ tablespoon) every 1 - 3 years to check the status of your disease. An ECG will be repeated around Day 5, and then at about 6 weeks and about 3 months.

You will be asked to visit the doctor for a physical exam and to have vital signs measured periodically. These visits will be scheduled at least every 3 to 4 months the first year. After the first year, the study staff will recommend that you have physical exams once every year. The visits may be scheduled more often depending on the status of the disease.

Treatment may be continued for up to 8-10 years or as long as the doctor feels it is necessary to control the leukemia. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

This is an investigational study. Nilotinib is FDA approved. A total of 150 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Ph-positive or Bcr-positive CML in early chronic phase CML (i.e., time from diagnosis 12 months). Except for hydroxyurea, patients must have received no or minimal prior therapy, defined as <1 month (30 days) of prior interferon-alpha (with or without cytarabine) and/or an FDA-approved Tyrosine Kinase Inhibitor (TKI). Patients with de novo accelerated phase will be treated but analyzed separately.
2. Age >/= 16 years (Age >18 years to participate in optional symptom burden assessment)
3. Eastern Cooperative Oncology (ECOG) performance of 0-2.
4. Adequate end organ function, defined as the following: total bilirubin < 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT/SGPT) < 2.5 x ULN, creatinine < 1.5 x ULN.
5. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
6. Reliable telephone access to receive calls from an interactive voice response system (IVR) (only applicable to patients who will participate in optional symptom burden assessment).

Exclusion Criteria:

1. New York Heart Association (NYHA) cardiac class 3-4 heart disease as well as impaired cardiac function defined as: left ventricular ejection fraction (LVEF) < 45% as determined by Multigated Acquisition Scan (MUGA) scan or electrocardiogram; Complete left bundle branch block; Use of cardiac pacemaker; ST depression of > 1 mm in 2 or more leads and/or T wave inversions in 2 or more continuous leads; Congenital long QT syndrome; History of, or presence of significant ventricular or atrial tachyarrhythmia's; Clinically significant resting bradycardia (< 50 bpm); QTc > 450 msec on screening ECG (using the QTcF formula);
2. (Continued from #1) Right bundle branch block plus left anterior hemiblock, bivascular block; Myocardial infarction within 12 months prior to starting AMN107; Unstable angina diagnosed or treated within the past 12 months; Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
3. Patients with active, uncontrolled psychiatric disorders including: psychosis, major depression, and bipolar disorders.
4. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Surgical sterilization is considered non-childbearing potential. Female patients of reproductive potential must agree to employ an effective method of birth control (hormonal or barrier) throughout the study and for up to 3 months following discontinuation of study drug.
5. Patients with severe and/or uncontrolled medial disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection [persistent fever and worsening clinical condition]).
6. Patient with known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
7. Patient with known diagnosis of human immunodeficiency virus (HIV) infection.
8. Patients in late chronic phase (i.e., time from diagnosis to treatment >12 months) or blastic phase are excluded. The definitions of CML phases are as follows: A. Early chronic phase: time from diagnosis to therapy < 12 months Late chronic phase: time from diagnosis to therapy > 12 months.B. Blastic phase: presence of 30% blasts or more in the peripheral blood or bone marrow. C. Accelerated phase CML: presence of any of the following features: * Peripheral or marrow blasts 15% or more.
9. (Cont. #8)Peripheral or marrow basophils 20% or more. *Thrombocytopenia < 100 x 10(9)/L unrelated to therapy. * Documented extramedullary blastic disease outside liver or spleen due to past causes D. Clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph chromosome is part of accelerated phase CML. Ph chromosome variants or complex Ph chromosome translocations are not considered to indicate disease acceleration.
10. ( Cont # 8) We have recently found clonal evolution to have a variable prognostic impact and may be suppressed with Interferon therapy (IFN-a therapy). Hence these patients, like others with de novo accelerated phase, will be eligible, and analyzed separately.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-06-27 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Kantarjian H, Boddu PC, Nogueras-Gonzalez GM, Verstovsek S, Garcia-Manero G, Borthakur G, Sasaki K, Kadia TM, Sam P, Ahaneku H, O'Brien S, Estrov Z, Ravandi F, Jabbour E, Cortes JE. Analysis of cardiovascular and arteriothrombotic adverse events in chronic-phase CML patients after frontline TKIs. Blood Adv. 2019 Mar 26;3(6):851-861. doi: 10.1182/bloodadvances.2018025874. PMID 30885996
- [Derived] Issa GC, Kantarjian HM, Gonzalez GN, Borthakur G, Tang G, Wierda W, Sasaki K, Short NJ, Ravandi F, Kadia T, Patel K, Luthra R, Ferrajoli A, Garcia-Manero G, Rios MB, Dellasala S, Jabbour E, Cortes JE. Clonal chromosomal abnormalities appearing in Philadelphia chromosome-negative metaphases during CML treatment. Blood. 2017 Nov 9;130(19):2084-2091. doi: 10.1182/blood-2017-07-792143. Epub 2017 Aug 23. PMID 28835440
- [Derived] Jain P, Kantarjian H, Nazha A, O'Brien S, Jabbour E, Romo CG, Pierce S, Cardenas-Turanzas M, Verstovsek S, Borthakur G, Ravandi F, Quintas-Cardama A, Cortes J. Early responses predict better outcomes in patients with newly diagnosed chronic myeloid leukemia: results with four tyrosine kinase inhibitor modalities. Blood. 2013 Jun 13;121(24):4867-74. doi: 10.1182/blood-2013-03-490128. Epub 2013 Apr 25. PMID 23620574
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib
Started | 148
Completed | 148
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 124
  >=65 years | 21
Age, Continuous [Median (Full Range); unit: years] | 51 [17 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 134
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 148

OUTCOME MEASURES:

1. Primary Outcome: Participants With Complete Molecular Response (Molecular CR)
Description: Polymerase chain reaction (PCR) Ratio BCR-Abl/Abl of 0% after 12 months of therapy with Nilotinib by international standard.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 148
Participants | 23

2. Secondary Outcome: Number of Participants With Complete Cytogenetic Response (CCyR)
Description: Complete hematologic remission classified according to suppression of Philadelphia chromosome (Ph) by cytogenetics or i Fluorescence in situ hybridization (FISH)
  1. No cytogenetic response - Ph positive 100%
  2. Minor cytogenetic response - Ph positive 35-90%
  3. Partial cytogenetic response - Ph positive 1-34%
  4. Complete cytogenetic response - Ph positive 0% Major cytogenetic response = complete + partial (Ph positive <35%)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 148
Participants | 131

ADVERSE EVENTS:
Time Frame: Up to 11.5 years
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 7/148
Serious Adverse Events (participants affected / at risk) | 47/148
Other Adverse Events (participants affected / at risk) | 148/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib (N=148)
Left Buccal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac Chest Pain (Cardiac disorders) | 6 (7)
Cardiac ischemia/infarction (Cardiac disorders) | 5 (6)
CNS Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
CNS Ischemia (Nervous system disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Elevated Creatinine (Investigations) | 1 (1)
Death (General disorders) | 2 (2)
Revision right hip arthroplasty (Surgical and medical procedures) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Flu like Syndrome (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (3)
GI Pain (Gastrointestinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Hysterectomy (Surgical and medical procedures) | 2 (2)
Knee Replacement (Surgical and medical procedures) | 1 (1)
Pain (General disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urethra Stricture (Renal and urinary disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Valvular heart disease (Cardiac disorders) | 1 (2)
Vascular Stenosis (Vascular disorders) | 1 (1)
Abdoninal Pain (Gastrointestinal disorders) | 8 (9)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Angioplasty with Stent Placement (Surgical and medical procedures) | 1 (1)
Back Pain (General disorders) | 2 (2)
Cholecyctitis (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hip Replacement (Surgical and medical procedures) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Elevated Transaminases (Investigations) | 1 (1)
Infection (Infections and infestations) | 3 (4)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3)
Neoplasm squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Persomality/behavioral -alcohol treatment (Psychiatric disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Psychosis (Psychiatric disorders) | 1 (1)
Secondary Malignancy - Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib (N=148)
Rash (Skin and subcutaneous tissue disorders) | 76 (76)
Fatigue (General disorders) | 65 (65)
Elevated bilirubin (Investigations) | 84 (84)
Elevated Aminotransferases (Investigations) | 71 (71)
Hypertension (Vascular disorders) | 26 (30)
Cardiovascular Ischemia (Cardiac disorders) | 11 (11)
Arrhythmia (Cardiac disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT00129740/Prot_SAP_000.pdf